CLINICAL TRIAL: NCT01757249
Title: A Single Centre Open-label Randomised Controlled Trial of Long Term Pituitary Down-regulation Before in Vitro Fertilisation for Women With Endometriosis: a Pilot Study
Brief Title: Pituitary Down-regulation Before IVF for Women With Endometriosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit sufficient participants
Sponsor: University of Oxford (Other)
Collaborators: Oxford Fertility Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDOG-12/SC/0645; 2012-004954-27 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Fertility
MeSH Terms: interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 OCP (Experimental): Combined oral contraceptive pill (OCP) (Microgynon 30) containing Levonorgestrel/Ethinylestradiol 150/30mcg. Taken orally on a continuous regime for 8 weeks, once a day.
  Interventions: Drug: Combined Oral Contraceptive Pill (Microgynon 30)
- Group 2 Control (No Intervention): Control Group - no intervention

INTERVENTIONS:
Drug: Combined Oral Contraceptive Pill (Microgynon 30) — Pre-IVF treatment for 8 weeks
  Other Names: Microgynon 30
  Arms: Group 1 OCP

SUMMARY:
Endometriosis is a hormone dependent disease of women, in which endometrial tissue (the cells which line the uterus or womb) are found outside the uterus (womb). Some women with endometriosis may be infertile. However, treatments for infertility such as in vitro fertilization (IVF) or IVF with intracytoplasmic sperm injection (IVF-ICSI) appear to be less successful, i.e. the pregnancy rates are lower, for women with endometriosis than for women who may be infertile for other reasons.

Since endometriosis is hormone dependent, it has been suggested that suppressing the activity of hormones produced by the ovaries (which affect endometrial growth) may inactivate endometriosis and so increase the chances of pregnancy. Recently it has been proposed that taking the oral contraceptive pill (OCP) for 6 to 8 weeks before IVF or IVF-ICSI treatment could be used for this purpose.

For our study, which is a randomised controlled trial, women with endometriosis meeting the study criteria planning to undergo IVF or IVF-ICSI at the Oxford Fertility Unit will be recruited. Study participants will be randomised into 2 arms: experimental group and control group. The experimental group will be instructed to complete an 8 week course of OCP before beginning standard IVF treatment. The control group do not take any study medication before beginning standard IVF treatment. The IVF or IVF-ICSI treatment for both groups is not altered by participation in the study.

The aim of the study will be to determine if pretreatment with OCP improves IVF or IVF-ICSI success rates, such as live birth and pregnancy rates, in patients who suffer from endometriosis. The study is funded by the Oxford Fertility Unit.

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent for participation in the study.

* Female aged 18 to 39 years old.
* Intending to undergo treatment with a first, second or third cycle of IVF or IVF-ICSI.
* Diagnosed with any degree of endometriosis or endometrioma.
* Participants must meet World Health Organisation Group 1 or 2 eligibility requirements for Combined Oral Contraceptive use.

Exclusion Criteria:

The participant does not understand the English language, or has special communication needs. This is because it is impractical to provide, for this small scale study, information sheets and consent forms in other languages except English.

* The patient has already undergone 3 or more IVF or IVF-ICSI cycles.
* Patients who are already taking any medication to treat endometriosis such as progestins, OCP, Gonadotrophin Releasing Hormone agonists, danazol, mirena, etc. or who have done so within the last 3 months.
* Participants who do not meet World Health Organisation Group 1 or 2 eligibility requirements for Combined Oral Contraceptive use.

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Live birth rate | up to 40 weeks following embryo transfer date
  The birth of a live child after 24 gestational weeks

SECONDARY OUTCOMES:
IVF Cycle outcomes | up to 40 weeks following embryo transfer date
  Cancelled cycles, failed cycles - negative pregnancy test, biochemical pregnancy, clinical pregnancy, miscarriage, stillbirth
Treatment responses per cycle | up to one week after egg collection
  No. of follicles aspirated, No. of oocytes retrieved, No. of cleavage embryos obtained, Total dose and duration of Gonadotrophins
Number of cases of Ovarian Hyperstimulation Syndrome | Up to 4 weeks after final embryo transfer
Multiple pregnancy rate | Up to 6 weeks after final embryo transfer
Number of ectopic pregnancies | up to 6 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Tim Child, Principal Investigator — University of Oxford
Locations (1):
- NDOG, University of Oxford, Oxford, United Kingdom